CLINICAL TRIAL: NCT01538667
Title: Non-blinded, Single Dose, Single Centre Trial to Assess the Pulmonary Deposition as Well as Pharmacokinetics, Safety and Tolerability of 99mTc Labeled Ciprofloxacin When Delivered as a Single Dose From a Dry Powder Inhaler to Healthy Subjects With and Without Charcoal Block and Patients Suffering From Bronchiectasis and COPD
Brief Title: Study to Characterize Lung Deposition, Pharmacokinetics, Safety and Tolerability of Single Inhalations of Radiolabeled Ciprofloxacin Dry Powder in Healthy Subjects and Patients With Chronic Lung Diseases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11523; 2011-000342-38 (EudraCT Number)
Record Dates: First submitted 2012-02-21; First posted 2012-02-24 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Respiratory System
Keywords: Lung; Scintigraphy; Pharmacokinetics; Inhalation; Ciprofloxacin
MeSH Terms: conditions — Respiratory Aspiration | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: Ciprofloxacin (Cipro Inhale, BAYQ3939)
- Arm 2 (Experimental)
  Interventions: Drug: Ciprofloxacin (Cipro Inhale, BAYQ3939)
- Arm 3 (Experimental)
  Interventions: Drug: Ciprofloxacin (Cipro Inhale, BAYQ3939)
- Arm 4 (Experimental)
  Interventions: Drug: Ciprofloxacin (Cipro Inhale, BAYQ3939)

INTERVENTIONS:
Drug: Ciprofloxacin (Cipro Inhale, BAYQ3939) — 50 mg single powder dose of 99mTc labeled ciprofloxacin PulmoSphere inhalation powder inhaled by healthy subjects
  Arms: Arm 1
Drug: Ciprofloxacin (Cipro Inhale, BAYQ3939) — 50 mg single powder dose of 99mTc labeled ciprofloxacin PulmoSphere inhalation powder inhaled by healthy subjects under charcoal block
  Arms: Arm 2
Drug: Ciprofloxacin (Cipro Inhale, BAYQ3939) — 50 mg single powder dose of 99mTc labeled ciprofloxacin PulmoSphere inhalation powder inhaled by COPD patients
  Arms: Arm 3
Drug: Ciprofloxacin (Cipro Inhale, BAYQ3939) — 50 mg single powder dose of 99mTc labeled ciprofloxacin PulmoSphere inhalation powder inhaled by bronchiectasis patients
  Arms: Arm 4

SUMMARY:
The purpose of this study is to characterize variability and extent of the deposition of ciprofloxacin in the respiratory tract of healthy subjects in comparison to patients with chronic lung diseases after inhalation of a single 50 mg dry powder dose containing 32 mg active substance. In addition the safety and pharmacokinetics of ciprofloxacin will be evaluated. In this study the radiolabeled substance will be administered and scintigraphy imaging techniques will be used to demonstrate the lung deposition visually. In the healthy subjects an additional pharmacokinetic method is used to calculate lung deposition indirectly based on pharmacokinetic data derived from plasma. For this purpose they will inhale at a separate occasion another dose of ciprofloxacin after having ingested activated charcoal. The latter serves to bind ciprofloxacin which is swallowed down during the inhalation maneuver in the gastrointestinal (GI) tract, thus preventing its uptake into the blood (charcoal block). Safety investigations will focus on local tolerability in the lung.

Pharmacokinetics is to see how the body absorbs, distributes, breaks down and gets rid of the study drug.

Results from this study will be used to show how the drug is distributed in the human lung.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for all subjects:

  * Understanding of the study and written informed consent prior to any study-related procedures
* Additional inclusion criteria for healthy subjects:

  * Age: 18 to 65 years (inclusive) at screening visit
  * Males
  * Non- or ex-smokers who smoked < 5 pack-years and stopped smoking > 1 year prior to screening visit
  * Results of laboratory tests within the normal ranges; minor deviations are acceptable provided that they are not judged clinically significant by the investigator
* Additional inclusion criteria for patients with COPD (chronic obstructive pulmonary disease):

  * Age: 40 to 70 years (inclusive) at screening visit
  * Males and females
  * All patients must have a diagnosis of COPD of Stage II or III according to the GOLD (Global Initiative for Chronic Obstructive Lung Disease) Classification (post-bronchodilator forced expiratory volume in 1 second (FEV1): 80% > FEV1 ≥ 30% of predicted values and a post-bronchodilator FEV1/FVC ≤ 70% (FVC = forced vital capacity)
  * Minimum smoking history of 10 pack-years
* Additional inclusion criteria for patients with bronchiectasis:

  * Age: 18 to 75 years (inclusive) at screening visit
  * Males and females
  * Diagnosis of bronchiectasis

Exclusion Criteria:

* Known hypersensitivity, allergy or intolerance to study drug formulation ingredients
* Febrile illness within 1 week prior to screening visit
* Concomitant severe diseases (judged by the investigator) or diseases which are contraindications for the use of inhaled ciprofloxacin
* Use of ciprofloxacin within 30 days before screening visit
* Use of systemic or topical medicines or substances which oppose the study objectives or which might influence them, e.g. systemic administration of antibiotics which are subject to renal excretion (e.g. beta-lactam antibiotics, levofloxacin, ofloxacin, etc.), furosemide and antacids
* Donation of more than 450 mL of blood within 4 weeks before screening visit
* Clinically relevant findings in the ECG
* Clinically relevant abnormal laboratory values suggesting an unknown disease and requiring further clinical investigation
* Participation in another clinical study less than 8 weeks prior to screening visit
* Pulmonary exacerbation within the 6 weeks prior to screening
* History of lung transplant or any lung surgery or on any thoracic surgery waiting list
* Additional exclusion criteria for healthy subjects

  * Lung function measurements outside normal limits (Normal values: FEV1/FVC > 70% and FEV1 and FVC > 80% of predicted)
* Additional exclusion criteria for patients

  * Regular use of daytime oxygen therapy
  * Diagnosis of bronchial asthma
  * Diagnosis of clinically evident bronchiectasis (COPD patients)
  * Total blood eosinophil count >/= 600/mm3.
  * Completion of a pulmonary rehabilitation program in the six weeks prior to screening visit or current participation in a pulmonary rehabilitation program
  * Change in dose or type of any medications within 4 weeks prior to the screening visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Ciprofloxacin pharmacokinetics including lung deposition | Within 24 hours after treatment
  Firstly, scintigraphic imaging, a non-invasive method using a radioactive (99mTc-) label tagged to the formulation, will be used to describe the distribution and deposition of a single inhaled dose of Ciprofloxacin Dry Powder Inhalation (DPI) in the lung quantitatively. Secondly, based on blood sampling over a period of 24 hours after inhalation non-compartmental pharmacokinetic parameters of ciprofloxacin will be calculated to determine the systemic exposure to drug following inhalation of a single 32.5 mg Ciprofloxacin dose.

SECONDARY OUTCOMES:
Adverse Events collection | Within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Gauting, Bavaria, Germany